CLINICAL TRIAL: NCT04872192
Title: Evaluation of the Analgesic Efficacy of Bilateral Ultrasound-guided Transversus Thoracic Muscle Plane Block on Post-sternotomy Pain: a Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Transversus Thoracic Muscle Plane Block on Post-sternotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, assistant professor of anaesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 20/ 2020/ 2021
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
Keywords: transversus thoracic muscle block; adults; cardiac surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus (Active Comparator): patients received transversus thoracic muscle plane block and injection of 15 ml bupivacaine 0.25% on each side.
  Interventions: Other: transversus thoracic muscle plane block
- general anaesthesia group (Sham Comparator): the same bilateral technique was done on both sides and 15 ml saline was injected during each side of TTPB technique.
  Interventions: Other: general anaesthesia

INTERVENTIONS:
Other: transversus thoracic muscle plane block — transversus thoracic muscle plane block by injection of 15 ml of bupivacaine 0.25% on each side combined with general anaesthesia
  Arms: transversus
Other: general anaesthesia — transversus thoracic muscle plane block by injection of 15 ml of saline on each side combined with general anaesthesia
  Arms: general anaesthesia group

SUMMARY:
Patients were randomly allocated to either Tansversus group (T group) and general anesthesia (N group).Patient demographic data, preoperative medical status, left ventricular function, and operative data (total ischemic time, number of grafts) were recorded. The primary outcome of the study was Percentage of patients needed additional doses of morphine . The secondary outcomes included postoperative visual analogue pain scores performed after patient extubation for pain assessment at rest (0 = no pain, 10 = maximum unbearable pain) at time of extubation, 8h, 12 h,18 h and 24 hours postoperatively were recorded, when pain score >4, patients were given morphine 0.05 mg/kg administered by a physician who was blinded to the nature of the study, time needed for first rescue analgesic, postoperative blood pressure and heart rate were recorded immediately on admission then 2 hours, 4 hours, 6 hours, 12 and 24 hours postoperatively, in addition to extubation time, length of ICU stay, the incidence of complications related to the technique such as hemothorax or pneumothorax, arrhythmias, and local anesthetic toxicity were recorded. The end-point was difficult weaning from cardiopulmonary bypass, major postoperative bleeding which required re-exploration or allergy to any agents needed for anesthesia. All complications were managed according to surgical and medical guidelines.

DETAILED DESCRIPTION:
Patients were randomly allocated to either Tansversus group (T group) and general anesthesia (N group). The patients were randomized using a computer-generated random number in various block sizes in 1:1 ratio. Randomisation was done using the SAS statistical package version 9.3 (SAS institute, Cary, NC, USA) by a statistician who was not involved in the study.

In the Tansversus group (n=30), prior to surgical incision, a 12 L-RS linear probe of the Sonosite M Turbo ultrasound system (National electrical manufacturers, USA). Probe was put beneath the clavicle next to the sternal edge and the second rib was visualized. Sliding the probe on the ribs downward till reaching the fifth rib. The probe was rotated 90 degrees and placed in the fouth intercostal space between the fourth and fifth ribs at the edge of the sternum. A 20-gauge Tuohy needle was introduced from lateral-to-medial in the plane between the internal intercostal muscles IIM and the transversus thoracic muscle TTM. Injection of 1 mL of normal saline was done to identify this plane followed by injection of 15 ml bupivacaine 0.25% on each side and observation of the local anesthetic spread, and pushing on the pleura confirmed the correct injection of the local anesthetic. This technique was done on the other side. It is important to identify the internal mammary artery IMA which was visualized as a hypoechoic pulsatile structure to avoid inadvertent puncture of the artery and subsequent bleeding and proper visualization of the IMA can facilitate the block. In N group (n=30), the same bilateral technique was done on both sides and 15 ml saline was injected during each side of TTPB technique. All the blocks were done by a single experienced anesthetist. Drug packs were prepared before commencement of the study by a pharmacist who was unaware of the nature of the study Hemodynamic changes, such as high blood pressure or significant tachycardia, additional 0.5- to-1 micrograms/kg IV doses of fentanyl were administered.

Median sternotomy was performed in all cardiac surgical procedures. At the end of the cardiac surgical procedure, all patients were transferred to the ICU after surgery to maintain the hemodynamics, warming them up with control of bleeding and correction of hemoglobin level, serum electrolytes and acid-base balance. A standard postoperative analgesia was accomplished by acetaminophen 1 gm/6 hours.The protocol for postoperative care was implemented for all patients by well-trained, qualified bedside nurses supervised 1:1 by well-trained ICU consultants. All patients were extubated when deemed clinically appropriate according to the local ICU protocol, by ICU staff, when the patient was able to maintain spontaneous breathing after extubation. The patients were encouraged to sit on a chair and mobilize with the assistance of health care providers in the ICU then the physiotherapist became responsible for improving mobility and rehabilitation of the patients till discharge from the hospital.

Patient demographic data, preoperative medical status, left ventricular function, and operative data (total ischemic time, number of grafts) were recorded. The primary outcome of the study was Percentage of patients needed additional doses of morphine The secondary outcomes included total dose of morphine requirements, postoperative visual analogue pain scores performed after patient extubation for pain assessment at rest (0 = no pain, 10 = maximum unbearable pain) at time of extubation, 8h, 12 h,18 h and 24 hours postoperatively were recorded, when pain score >4, patients were given morphine 0.05 mg/kg administered by a physician who was blinded to the nature of the study, time needed for first rescue analgesic, postoperative blood pressure and heart rate were recorded immediately on admission then 2 hours, 4 hours, 6 hours, 12 and 24 hours postoperatively, in addition to extubation time, length of ICU stay, the incidence of complications related to the technique such as hemothorax or pneumothorax, arrhythmias, and local anesthetic toxicity were recorded. The end-point was difficult weaning from cardiopulmonary bypass, major postoperative bleeding which required re-exploration or allergy to any agents needed for anesthesia. All complications were managed according to surgical and medical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* age between 55-74 years
* ASA II-III
* BMI<30

Exclusion Criteria:

* patients who were preoperatively intubated for more than 24 hours
* patients with complex cardiac procedures
* patient inability to communicate patients with severe pulmonary hypertension in addition to any contraindication to regional anesthesia

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients needed additional doses of morphine | 24 hours postoperative
  number of patients requiring additional doses of morphine

SECONDARY OUTCOMES:
postoperative visual analogue pain scores | time of extubation, 8 hours, 12 hours,18 hours and 24 hours postoperatively
  pain assessment at rest (0 = no pain, 10 = maximum unbearable pain)
postoperative total morphine dose | 24 hours postoperative
  dose of postoperative rescue morphine requirements

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Shokri, Principal Investigator — Ain Shams University; Ihab Ali, Study Director — AinShams university
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 4 months
Access Criteria: The collected data are coded, tabulated, and statistically analyzed using statistical package for social sciences software, version 17.0 (SPSS Inc., Chicago, Illinois, USA). Descriptive statistics are carried out for numerical parametric data and presented as mean±SD, whereas categorical data are presented as number and percentage. Variables such as demographic data and comorbidities are compared using the χ2-test. A P value less than 0.05 was considered significant.